CLINICAL TRIAL: NCT04813536
Title: Effect of Work Shift on the Nurses' Health in the Main Assiut University Hospital
Brief Title: Shift Work Health Effects
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Roshdy Elkhayat, lecturer, Assiut University
Other Study IDs: shift work
Record Dates: First submitted 2021-03-20; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Shift-work Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- nurses in Assiut university hospitals: currently working nurses exposed to shift work
  Interventions: Other: the Standard Shiftwork Index questionnaire; Other: complete blood picture; Other: lipid profile
- control group: currently working nurses not exposed to shift work
  Interventions: Other: the Standard Shiftwork Index questionnaire; Other: complete blood picture; Other: lipid profile

INTERVENTIONS:
Other: the Standard Shiftwork Index questionnaire — 1. Biographical information: This includes personal data (e.g., age, sex, marital status, and domestic situations), shift details (e.g., shift start and end times), organization of shiftwork, and general job satisfaction
  2. Sleep and fatigue: Measures the effect of shiftwork on perceived sleep quality and quantity and fatigue
Other: complete blood picture — 5ml blood to estimate changes of total leucocytic count, Hemoglobin, eosinophilic, monocyte
Other: lipid profile — 5ml blood to estimate changes of plasma triglycerides, total cholesterol, low-density lipoprotein cholesterol (LDL-C), and HDL-C

SUMMARY:
To identify the health effects of shift work on nurses in Assuit university hospitals .

To estimate effect of shift work on co-morbidities among nurses . To determine the shift work associated risk factors predisposing nurses to poor health outcomes and injuries.

DETAILED DESCRIPTION:
The word 'shiftwork' is commonly used to describe irregular, odd, untraditional working hours, or working hours that are away from day work period. Shiftwork dates back to the late 1800s, as applied to guardians of old kingdoms and in the military services. After the innovation of the light, shift work expanded for nonstop production as in steel factories, iron foundries, and material plants. Approximately one-fourth of the workforce in hospitals works unusual hours (away from the traditional diurnal work period) . Shiftwork has a number of advantages and disadvantages to employers, employees, and their families. The advantages for employers include optimal use of energy, facilities, and other resources through extended capital operating time. The advantages for employees include increased income, more free time for daily activities, and saving time by avoiding traffic rush hours. Shiftwork is associated with both short-term and long-term disadvantages on physical and psychophysiological health. Short-term effects include fatigue and difficulties with sleep. Difficulties with sleep are found to be the most common complaint among shift workers. Sleep disturbances were the main reasons that led shift workers to leave night shiftwork owing to disturbed health habits compared with day workers .Gastrointestinal disorders were reported 2-5 times more commonly among shift workers than daytime workers. These disorders range from minor complaints (e.g., constipation, heart burn, distension, and disturbed appetite) to serious gastrointestinal disorders, which may develop into chronic diseases such as chronic gastritis or peptic ulcers. Shiftwork has been also linked to type 2 diabetes and obesity as sleep deprivation activates the immune system and influences glucose metabolism .

An association between shiftwork and cardiovascular diseases (CVDs) has been reported. There is a higher risk for CVD such as hypertension, subclinical atherosclerosis, and ischemic heart disease compared with daytime workers . Different types of cancer have been reported in shift workers including cancers of the breast, colon, and endometrium. Shiftwork system causes circadian rhythm disruption, which is probably carcinogenic to humans.

Also, shiftwork causes disruption in both social and domestic lifestyle, which is a major consequence of shiftwork, especially with maternal employment that may have some adverse influences on their young children's cognitive and behavioral outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Active working nurses working in Assiut University Hospitals with minimum exposure to work shift for 1 year .
* Had free pre-employment records

Exclusion Criteria:

* Nurses don't record shift work exposure.
* Nurses with less than 1 year exposure to shift work, or don't recorded shift work exposure.
* Nurses known to had autoimmune disorder or endocrinal disorder before joining job.

Ages: 18 Years to 60 Years | Sex: Female
Age Groups: Adult
Study Population: Active working nurses working in Assiut University Hospitals with minimum exposure to work shift for 1 year
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
complete blood picture | once baseline at time of the data collection of study
  total leucocytic count
complete blood picture | once baseline at time of the data collection of study
  Hemoglobin
complete blood picture | once baseline at time of the data collection of study
  eosinophilic count
complete blood picture | once baseline at time of the data collection of study
  monocyte count
lipid profile | once baseline at time of data collection
  plasma triglycerides
lipid profile | once baseline at time of data collection
  total cholesterol
lipid profile | once baseline at time of data collection
  low-density lipoprotein cholesterol (LDL-C)
lipid profile | once baseline at time of data collection
  HDL-C
Sleep Questionnaire | once baseline at time of data collection
  part of standard shift work index,consists of 11 items and aims to identify sleep habits, as well as the extent to which sleep is depending on which shift has been or is about to be worked. A higher score is associated being associated with higher sleep disturbance

REFERENCES:
- [Background] Gadallah M, Hakim SA, Mohsen A, Eldin WS. Association of rotating night shift with lipid profile among nurses in an Egyptian tertiary university hospital. East Mediterr Health J. 2017 Jun 14;23(4):295-302. doi: 10.26719/2017.23.4.295. PMID 28634980
- [Background] Merchaoui I, Bouzgarrou L, Mnasri A, Mghanem M, Akrout M, Malchaire J, Chaari N. Influence of shift work on the physical work capacity of Tunisian nurses: a cross-sectional study in two university hospitals. Pan Afr Med J. 2017 Feb 2;26:59. doi: 10.11604/pamj.2017.26.59.11279. eCollection 2017. PMID 28451036
- [Background] Ferri P, Guadi M, Marcheselli L, Balduzzi S, Magnani D, Di Lorenzo R. The impact of shift work on the psychological and physical health of nurses in a general hospital: a comparison between rotating night shifts and day shifts. Risk Manag Healthc Policy. 2016 Sep 14;9:203-211. doi: 10.2147/RMHP.S115326. eCollection 2016. PMID 27695372
- [Background] Dehring T, von Treuer K, Redley B. The impact of shift work and organisational climate on nurse health: a cross-sectional study. BMC Health Serv Res. 2018 Jul 27;18(1):586. doi: 10.1186/s12913-018-3402-5. PMID 30053871